CLINICAL TRIAL: NCT06617689
Title: Effekt av Pasientundervisning på Drikkevaner og Munnhygiene Hos Pasienter Som gjennomgår Fedmekirurgi
Brief Title: Effect of Patient Education on Drinking Behaviour and Oral Hygiene in Patients Undergoing Bariatric Surgery
Acronym: BAR-VANNTANN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Helse Møre og Romsdal Hospital Trust (Unknown); Helse Nord-Trøndelag HF (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 705887
Record Dates: First submitted 2024-09-26; First posted 2024-09-27 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Obesity; Oral health
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Group-based teaching (Experimental): In this arm, all three educational activities are included: Teaching (in a group), distribution of free dental hygiene samples, and advice on reading the customised website. This arm is compared to Arm 2.
  Interventions: Other: Various levels of patient education
- Arm 2: Comparator to Arm 1 (Active Comparator): In this arm, patients are distributed free dental hygiene samples, and given advice on reading the customised website. This arm is compared to Arm 1.
  Interventions: Other: Various levels of patient education
- Arm 3: Goodiebag (Experimental): In this arm, patients are distributed free dental hygiene samples, and given advice on reading the customised website. This arm is compared to Arm 4.
  Interventions: Other: Various levels of patient education
- Arm 4: Comparator to Arm 3 (Active Comparator): In this arm, patients are adviced on reading the customised website. This arm is compared to Arm 3.
  Interventions: Other: Various levels of patient education

INTERVENTIONS:
Other: Various levels of patient education — The three interventions:
  GROUP BASED TEACHING In groups of 8-12 patients, 30 minutes of standardised teaching is given. The teaching focuses in particular on the changes in diet and the impact this has on oral pH, enamel erosion and caries; recommended oral hygiene; and good drinking habits.
  WEBSITE Website providing recommendations for oral hygiene and drinking habits, as well as in depth information on the topic.
  DENTAL HYGIENE SAMPLES These are samples relevant for maintaining proper oral hygiene, distributed free, together with a description of how to use them.

SUMMARY:
The background for the study is that many bariatric surgery patients struggle with their oral health after bariatric surgery. This is probably related to both physiological changes and changes in eating and drinking patterns. In addition, many have reduced oral health even before surgery, and a significant proportion also have dental treatment anxiety, which also affects their ability to seek dental treatment. In sum, this is probably a patient group that may be at risk of oral pathology.

Participants in the study will be randomly allocated to different patient education programmes. The three interventions are:

1. customised information on a website
2. education delivered by a clinician
3. distribution of free samples relevant to dental hygiene

The outcomes recorded are level of knowledge, drinking patterns, self-perceived oral health, and oral hygiene routines.

DETAILED DESCRIPTION:
Both caries and periodontitis are more prevalent among people with obesity. At the same time, we know that bariatric surgery is associated with poorer oral health expressed by caries, enamel erosion and short-term increased inflammation in the gums. Although we do not yet have evidence to determine causality, we suspect that oral health in bariatric surgery patients is further impaired by both systemic effects (hyposalivation, altered oral microbiome, reflux and vomiting) and by altered eating and drinking patterns after surgery (acid exposure with subsequent demineralisation of tooth enamel).

The patient's own diet and oral hygiene can be an opportunity to prevent or slow down such oral problems, but requires personal effort and must be a special focus in patient education.

Patient education is one of the hospital's statutory duties, but the quality of patient education is rarely systematically investigated. This project investigates the effect of three alternative educational interventions on patients' drinking habits, oral hygiene routines, knowledge level and oral health. The three interventions are a website with adapted patient information, group-based education given by healthcare professionals, and distribution of relevant product samples to maintain oral hygiene. Patients are randomised between the different educational interventions.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for bariatric surgery at a Norwegian hospital

Exclusion Criteria:

* Insufficient language skills
* Lack of consent competency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Drinking habits | Baseline to 6 months postop. to 24 months postop.
  Reported intake plain water with no additives

SECONDARY OUTCOMES:
Dental hygiene | Baseline to 6 months postop. to 24 months postop.
  Self-reported dental hygiene
Level of knowledge | Baseline to 6 months postop. to 24 months postop.
  Knowledge reflecting the central parts of the patient education

OTHER OUTCOMES:
Oral health | Baseline to 6 months postop. to 24 months postop.
  Self-reported oral health, including OHIP14

CONTACTS AND LOCATIONS:
Overall Officials: Magnus N Strømmen, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Patient education website in Norwegian, English and Polish — http://www.bar-oral.no